CLINICAL TRIAL: NCT05954793
Title: INNER-B-APAC - Asian Pacific Post-market Clinical Follow-up Study in Patients With Thoracoabdominal Aortic Aneurysms Treated With E-nside TAAA Multibranch Stent Graft System
Brief Title: A PMCF Study in Patients With Thoracoabdominal Aortic Aneurysms Treated With E-nside TAAA Multibranch Stent Graft System (INNER-B-APAC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: INNER-B-APAC
Record Dates: First submitted 2023-06-23; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Thoracoabdominal Aortic Aneurysm
Keywords: aneurysm; thoracoabdominal; aortic; vascular; surgery
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The INNER-B-APAC post-market clinical follow-up study is undertaken to demonstrate the safety and clinical performance of the E-nside TAAA Multibranch Stent Graft System used in endovascular treatment of patients with thoracoabdominal aortic aneurysms.

DETAILED DESCRIPTION:
In this study, patients will be observed who are planned to be treated an E-nside TAAA Multibranch Stent Graft System for endovascular repair of a degenerative, atherosclerotic thoracoabdominal aortic aneurysm. The E-nside TAAA Multibranch Stent Graft will be implanted at the discretion of the treating physician. Participating physicians will be asked to provide their observations collected during routine care for patients he/she had decided to treat with the E-nside TAAA Multibranch Stent Graft System. Informed consent of the patients to allow the use of their clinical records for the purpose of this observational study will be obtained before data are being collected. Patient data will be documented in an eCRF at the following time points: Pre-operative planning, intervention(s), discharge(s) from hospital, 30 days, 3-6 and 12 months follow-up. The period of data collection will be approximately 12 months (depending on the time point of the 12 months FU visit) from the index procedure for each patient. A 100% source data verification will be performed regarding patient information and consent, criteria of patients to be documented, pre-operative planning, intervention(s), treatment results, adverse events, death, and reintervention. Complete DICOM image files of the CT scans will be sent to a CoreLab for independent second evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 85 years old
* Patient has a degenerative, atherosclerotic thoracoabdominal aortic aneurysm
* Patient has adequate iliac/femoral access compatible with an 8.5 mm OD delivery system
* Patient's aorta has no distinct angulation in the thoracovisceral segment of the aorta ranging from 40 mm proximal to the celiac trunk to 20 mm distal to the lowest renal artery
* All target branch vessels are suitable for antegrade cannulation
* Diameter of the landing zone in each branch vessel to be treated is ≥ 5 mm
* Length of landing zone in each branch vessel to be treated is ≥ 15 mm (preferably ≥ 20 mm)
* Patient must be available for the appropriate follow-up times for the duration of the study
* Patient has signed the informed consent before implantation of the E-nside Stent Graft

Exclusion Criteria:

* Patient has allergies to materials necessary for endovascular repair (e.g. contrast media, anticoagulants or heparin, nitinol, polyester, gold, platinum-iridium)
* Patient has systemic infection or suspected systemic infection
* Patient has an infectious aneurysm
* Patient has an inflammatory aneurysm
* Patient has a ruptured aneurysm
* Patient has a traumatic aneurysm
* Patient has a symptomatic aneurysm
* Patient has an aortic dissection
* Patient has a congenital degenerative collagen disease or connective tissue disorder
* Diameter of ostium of branch vessel to be treated < 4 mm
* Patient has thrombocytopenia (platelet count < 150000/μl)
* Patient has an eGFR < 30 ml/min/1.73m2 before the intervention
* Patient has untreated hyperthyroidism
* Patient has a malignancy (progressive, stable or partial remission)
* Patient had a myocardial infarction or cerebrovascular accident < 3 months ago
* Patient is planned to be treated with a chimney in the left subclavian artery
* Patient has had a previous surgical repair of descending thoracic aorta
* Patient will be treated or had been treated with a Nellix (Endologix) or Ovation (Endologix) or Altura (Lombard Medical) or Anaconda (Vascutek) stent graft
* Patient is enrolled or plans to be enrolled in another clinical study
* Patient is pregnant or breastfeeding or planning to become pregnant during the course of the study.
* Patient has a life expectancy of less than 3 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with degenerative, atherosclerotic thoracoabdominal aortic aneurysm who are scheduled for implantation of an E-nside TAAA Multibranch Stent Graft at their physician's discretion and who are eligible in accordance with the criteria listed below.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Rate of all-cause mortality

SECONDARY OUTCOMES:
Mortality | 3-6 months, 12 months
  Rate of all-cause mortality
Rupture | through study completion, an average of 12 months
  Rate of patients with aneurysm rupture
Major adverse events | Prior to Discharge, 30 days, 3-6 months, 12 months
  Rate of patients with major adverse events
Number of interventions | Intra-Op
  Rate of interventions in peri-operative periods
Time E-nside delivery system remained in access vessels | through study completion, an average of 12 months
  Rate of time intervals the E-nside delivery system remained in the access vessels in relation to the number of branches treated with pre-cannulation
Reinterventions | 30 days, 3-6, 12 months
  Rate of reinterventions
Type Ia, Ib, Ic, II, III, IV endoleaks and endoleaks of unknown origin | 12 months
  Rate of patients with type Ia, Ib, Ic endoleak (at 12 months follow-up)
Intercomponent separation | Prior to Discharge, 30 days, 3-6 months, 12 months
  Rate of patients with intercomponent separation at the proximal or distal end of the E-nside stent graft > 10 mm
Loss of device integrity | Prior to Discharge, 30 days, 3-6 months, 12 months
  Rate of patients with loss of device integrity (stent fracture and tear in graft material and suture break)
Kinking of E-nside Stent Graft or bridging stents | Prior to Discharge, 30 days, 3-6 months, 12 months
  Rate of patients with E-nside stent graft or bridging stent kinking
Primary and secondary patency (overall and separately for each type of branch) | Prior to Discharge, 30 days, 3-6 months, 12 months
  Rate of primary/secondary patency of bridging stents Rate of primary/secondary patency of the bridging stent of the celiac trunk Rate of primary/secondary patency of the bridging stent of the superior mesenteric artery Rate of primary/secondary patency of the bridging stent of the right renal artery Rate of primary/secondary patency of the bridging stent of the left renal artery Rate of primary/secondary patency of branch vessels treated
Stent graft infection | through study completion, an average of 12 months
  Rate of patients with stent graft infection
Primary and secondary technical success | 24 hours
  Rate of patients with primary/secondary technical success
Primary and secondary clinical success | 12 months
  Rate of patients with primary/secondary clinical success
Stable, decreasing or increasing aneurysm size | 12 months
  Rate of patients with stable, decreasing or increasing aneurysm size
Removal or failure to implant the stent graft | through study completion, an average of 12 months
  Rate of patients with removal or failure to implant the E-nside TAAA Multibranch Stent Graft

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (4):
  - Alfred Health, Melbourne
  - Sir Charles Gairdner Hospital, Perth
  - Royal North Shore Hospital, Saint Leonards
  - Gold Coast University Hospital, Southport
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Waikato Hospital Hamilton, Hamilton
- Thailand (2):
  - Siriraj Hospital, Bangkok
  - Prince of Songkla University - Songklanagarind Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: No